CLINICAL TRIAL: NCT02200549
Title: Effects of Combined Cycle Training and Inspiratory Muscle Training on Exercise Performance ,Health-related Quality,Dyspnoea ,Body Composition,Depressive Symptomatology in Patients With Chronic Obstructive Pulmonary Disease(COPD)
Brief Title: Effects of Combined Cycle Training and Inspiratory Muscle Training in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX13902205193
Record Dates: First submitted 2014-07-20; First posted 2014-07-25 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: pulmonary rehabilitation; inspiratory muscle training; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Experimental): Neither cycle training nor inspiratory muscle training.
  Interventions: Device: Control group
- Cycle training group (Experimental): A 30-minute cycling training session is performed 3 days a week using calibrated cycle ergometer.
  Interventions: Device: calibrated cycle ergometer
- Combined group (Experimental): A 30-minute Combined training session is performed 3 days a week using calibrated cycle ergometer and threshold loading device.
  Interventions: Device: calibrated cycle ergometer and threshold loading device

INTERVENTIONS:
Device: Control group — Neither cycle training nor inspiratory muscle training.
  Arms: Control group
Device: calibrated cycle ergometer — The most common device to proform cycle training is calibrated cycle ergometer.
  Arms: Cycle training group
Device: calibrated cycle ergometer and threshold loading device — Combined cycle training and inspiratory muscle training.The threshold loading device is composed of a mouth -piece attached to a small plastic cylinder that contains a spring-loaded poppet value. The valve opens to permit inspiratory flow only once the person has generated adequate negative intrathoracic pressure to condense the spring.
  Arms: Combined group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) ，the fourth leading cause of death in the world, represents an important public health challenge. It is also a major cause of chronic morbidity, mortality and disability throughout the world, leading to a heavy social and economic burden. For a long time, treatment of COPD mainly focus on drug therapy. Recently, pulmonary rehabilitation is recognized as a core component of the management of individuals with chronic respiratory disease, which has been clearly demonstrated to reduce dyspnea, increase exercise capacity, and improve quality of life.

Exercise training, widely regarded as the cornerstone of pulmonary rehabilitation , is one of the best available means of improving muscle function in COPD.The most commonly form is cycle training. Inspiratory Muscle Training (IMT) as an adjunct to exercise training has an additional benefit on inspiratory muscle strength, endurance and exercise capacity in patient with COPD.

There is insufficient evidence demonstrate greater benefits from combined inspiratory muscle training and cycle training. This study will evaluate the effects of combined inspiratory muscle training and cycle training in patients with COPD.

DETAILED DESCRIPTION:
The patients with COPD will participate in a rehabilitation program for 8 weeks. Participants in the proposed study will be randomly programmed into one of three intervention groups:

1. Cycle training program alone (performing on calibrated stationary cycle ergometer).
2. Combined cycle training and inspiratory muscle training(performing on calibrated stationary cycle ergometer and threshold loading device).
3. Neither cycle training nor inspiratory muscle training.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 and 75 years of age were eligible if they met the following criteria:

  * moderate to severe airflow obstruction (30≤ Forced Expiratory Volume At One Second(FEV1) <80% predicted and Forced Expiratory Volume At One Second/Forced Vital Capacity(FEV1/FVC)<70%)
  * Complaints of dyspnea on exertion
  * Clinically stable condition
  * No participation in a pulmonary rehabilitation program in the last year.

Exclusion Criteria:

* Patients were excluded if they had evidence of asthma and/or had experienced a major exacerbation in the 2 months before enrollment
* Required home oxygen therapy or experienced oxyhemoglobin desaturation below 85% with exercise
* And/or had other health problems that would interfere with exercise.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Exercise Performance (composite outcome measure) | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Exercise performance tests include field walking tests and cycle ergometer tests.

SECONDARY OUTCOMES:
Health-related quality (composite outcome measure) | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Health-related quality is a component of the broader concept of quality of life and is defined as satisfaction with health.The St. George's Respiratory Questionnaire (SGRQ) and Chronic Respiratory Disease Questionnaire (CRQ）; and its self-reported version are the most widely used disease-specific questionnaires.
inspiratory muscle function (composite outcome measure) | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Currently, a variety of methods can be used to evaluate respiratory muscle function, including maximal inspiratory (PImax)，expiratory pressures(PEmax) and inspiratory muscle endurance.
Symptom Evaluation (composite outcome measure) | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Individuals with chronic respiratory disease often have symptoms such as dyspnea, fatigue, cough, weakness, sleeplessness,and psychological distress.Instruments for assessment of multiple symptoms include COPD Assessment Test (CAT) and Modified Medical British Research Council Scale(mMRC).

OTHER OUTCOMES:
Depression and anxiety evaluation | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Hospital Anxiety and Depression Scale (HADS) was found to perform well in assessing the symptom severity and caseness of anxiety disorders and depression in both somatic, psychiatric and primary care patients and in the general population.
Composite outcomes | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Among patients with COPD there is increasing interest in the use of multidimensional indices to characterize the severity of the disease and better predict outcomes.Arguably the most well-known of these indices is the BODE Index.
Body Composition Monitor | The groups will be assessed at baseline (time zero) and at the end of the training protocol (week 8)
  Body composition abnormalities are prevalent in COPD.Human body composition analyzer can detect various elements of human body and analyze human health status.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No